CLINICAL TRIAL: NCT00158314
Title: Cognitive Behavioral Treatment for Pathological Gambling
Brief Title: Cognitive Behavioral Therapy for Treatment of Pathological Gambling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Nancy Petry, PhD, University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH060417-01 (NIH); R01MH060417-01 (NIH); DATR A2-AIR
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Gambling
Keywords: Pathological gambling; Gambler's anonymous; Cognitive behavioral therapy; CBT
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Referral to Gamblers Anonymous
Behavioral: Cognitive behavioral therapy
Behavioral: Cognitive behavioral self-help manual

SUMMARY:
This study will determine the effectiveness and cost-effectiveness of three different treatment strategies in reducing gambling behaviors.

DETAILED DESCRIPTION:
The number of pathological gamblers in the United States is steadily growing, leading to significant financial, psychological, and public health consequences. However, studies examining the effectiveness of treatment interventions for pathological gamblers are limited. This study will compare the effectiveness of three different treatment strategies, including referral to Gambler's Anonymous (GA), a self-help manual, and cognitive behavioral therapy (CBT), in reducing gambling behaviors and other problems related to pathological gambling.

This study will last 8 weeks. Participants will be randomly assigned to one of three interventions. Group 1 participants will be referred to GA and 8 weeks of CBT, which focuses on teaching skills to help reduce gambling urges and develop alternative behaviors to gambling. Group 2 participants will be referred to GA and given an 8-week self-help manual. Group 3 participants will be referred to GA alone. Questionnaires will be used to assess participants' gambling behavior and any personal, legal, or health problems they may be experiencing. The questionnaires will be completed at study entry, study completion, and at 6- and 12-month follow-up visits.

Participants will be asked to identify at least one person who knows about their gambling problem and will have regular contact with them during the study and for at least 1 year This person will be interviewed at the beginning of the study, and at Months 2, 6 and 12. Researchers will ask contact persons about participants' gambling behaviors, personal relationships, legal problems, use of health care and mental health services, and how the participant can be contacted if he or she moves.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00118391

http://clinicaltrials.gov/show/NCT00618462

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pathological gambling
* 3 or more gambling episodes within 60 days prior to study entry

Exclusion Criteria:

* Inability to read English at the 5th grade level
* Uncontrolled psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231
Dates: Start 1998-03; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI) gambling severity scores
time spent gambling
days of non-gambling

SECONDARY OUTCOMES:
Psychiatric symptoms
psychosocial functioning

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M. Petry, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States